CLINICAL TRIAL: NCT01154387
Title: A Two Part, Phase 1/2, Safety, PK and PD Study of TOL101, an Anti-TCR Monoclonal Antibody for Prophylaxis of Acute Organ Rejection in Patients Receiving Renal Transplantation
Brief Title: Evaluating Safety and Efficacy of TOL101 Induction Versus Anti-Thymocyte Globulin to Prevent Kidney Transplant Rejection
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tolera Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTI-121
Record Dates: First submitted 2010-06-26; First posted 2010-06-30 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: End Stage Renal Disease; Renal Transplant
Keywords: Kidney; Renal; Transplant; Kidney Transplant; Kidney Failure; Induction; Monoclonal; Antibody; T cell; Anti-rejection; Immunosuppression
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency | interventions — Antilymphocyte Serum; thymoglobulin; TOL-101; Steroids; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Anti-Thymocyte Globulin (Active Comparator): Anti-Thymocyte Globulin induction as part of an immunosuppressive regimen that includes steroids, MMF, and tacrolimus.
  Interventions: Drug: Anti-Thymocyte Globulin; Drug: Steroids; Drug: Tacrolimus; Drug: Mycophenolate mofetil (MMF)
- TOL101 (Dose A) (Experimental): TOL101 induction as part of an immunosuppressive regimen that includes steroids, MMF, and tacrolimus.
  Interventions: Drug: TOL101; Drug: Steroids; Drug: Tacrolimus; Drug: Mycophenolate mofetil (MMF)
- TOL101 (Dose B) (Experimental): TOL101 induction as part of an immunosuppressive regimen that includes steroids, MMF, and tacrolimus.
  Interventions: Drug: TOL101; Drug: Steroids; Drug: Tacrolimus; Drug: Mycophenolate mofetil (MMF)

INTERVENTIONS:
Drug: Anti-Thymocyte Globulin — 1.5mg/kg IV on Day of Transplant and 1.0-1.5 mg/kg IV once daily for a minimum of 4.5mg/kg and a maximum of 7.5mg/kg total cumulative dose
  Other Names: Thymoglobulin
  Arms: Anti-Thymocyte Globulin
Drug: TOL101 — Potential Therapeutic Dose (PTD)-A (0.28-56 mg to be determined in Phase 1/Part A ) IV once daily x 6-10 doses starting on Day of Transplant
  Arms: TOL101 (Dose A)
Drug: TOL101 — Potential Therapeutic Dose (PTD)-B (0.28-56 mg to be determined in Phase 1/Part A ) IV once daily x 6-10 doses starting on Day of Transplant
  Arms: TOL101 (Dose B)
Drug: Steroids — IV methylprednisolone prior to first 3 doses of study drug; oral prednisone tapered to 5-10 mg over 6 months
Drug: Tacrolimus — Oral administration started by 6 days post-transplantation and continued for 6 months
Drug: Mycophenolate mofetil (MMF) — Oral administration started by Day 1 post-transplantation and continued for 6 months

SUMMARY:
Induction therapy with antibodies is administered during transplant surgery and for a short period of time following transplant surgery in an effort to render the immune system less able to mount an initial rejection response. In general, induction therapy is associated with better outcomes compared to the absence of induction therapy. However, currently used induction agents, some of which are not labeled or indicated for induction therapy in transplantation, have drawbacks related to long-term immune system suppression increasing susceptibility to opportunistic infections or malignancies, and other immune-mediated side effects.

An unmet medical need exists for a more specific approach to prevent acute organ rejection, without unnecessarily exposing the patient to non-specific or open-ended immune suppression, which may exacerbate the risks of infections and malignancies. TOL101 is a novel antibody that targets a very specific immune cell type that is critical in the acute organ rejection response. In this two-part study, TOL101 will be evaluated for the prophylaxis of acute organ rejection when used as part of an immunosuppressive regimen that includes steroids, MMF, and tacrolimus in first time kidney transplant recipients.

This study will test the hypothesis that a more specific approach (with TOL101) to prevention of acute organ rejection may provide similar or better efficacy than the currently used induction antibodies (such as Anti-Thymocyte Globulin or Thymoglobulin) while carrying fewer risks in terms of opportunistic infections, malignancies and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a primary renal transplant from a living or standard criteria cadaveric donor
* Male or female 18-60 years of age
* Recipient with a PRA < 20%

Exclusion Criteria:

* Previous solid organ transplant
* Recipient of HLA-identical kidney allograft transplant
* Recipient of an ABO incompatible donor kidney
* Known HIV infection or other major infection
* History of malignancy within 3 years (excluding treated basal cell or squamous cell carcinoma of the skin) prior to enrollment
* History of tuberculosis
* Recipient with cardiovascular disease
* Treatment with immunosuppressive medications within 1 month prior to enrollment
* Known or suspected allergy to mice
* Pregnant or lactating
* Unable or unwilling to participate in all required study activities for the duration of the study (6 months)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of ascending doses of TOL101 and the effectiveness of TOL101 to target and downregulate T cells in patients undergoing first renal transplantation | 6 months
  The following safety parameters will be monitored: Adverse events, standard laboratory safety evaluations (hematology and serum chemistries), symptom constellation indicating cytokine release syndrome, serum concentrations of cytokines and nitric oxide, malignancies, CMV viremia, BKV viremia, EBV viremia and other infections

SECONDARY OUTCOMES:
The effects of ascending doses of TOL101 on CD3+ T lymphocyte numbers and other immune cell subsets | 14 days post-transplant (Part A); 6 months (Part B)
The pharmacokinetic (PK) profile of TOL101 in renal transplant recipients and the exposure-response (PK parameter to CD3+ T lymphocyte numbers) relationship over time | 14 days post-transplant
Biopsy-proven acute organ rejection | 6 months
Graft survival | 6 months
Patient survival | 6 months
Renal function by measured GFR at 6 months post-transplant and urine protein to creatinine ratio at 3 and 6 months post-transplant | 6 months
Delayed graft function | first 7 days post-transplant
Immunogenicity of TOL101 by measurement of anti-TOL101 antibodies | at 14 and 28 days post-transplant
The presence of Donor Specific Antibody at 3 months (Part B only) and 6 months post-transplant | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Flechner, MD, Principal Investigator — The Cleveland Clinic
Locations (12):
- United States (12):
  - University of Colorado Denver, Aurora, Colorado
  - University of Kentucky, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - St Barnabas Medical Center, Livingston, New Jersey
  - Buffalo General Hospital, Buffalo, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - Baylor All Saints, Fort Worth, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia